CLINICAL TRIAL: NCT01141920
Title: Comparison of Two Different Counseling Schedules on Treatment Response of New Admissions to Methadone Maintenance
Brief Title: Comparison of Two Counseling Induction Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michael Kidorf, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: da012347-4
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Methadone; Drug Use Disorders
Keywords: treatment retention; methadone maintenance; treatment induction; Retention in methadone maintenance treatment
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3-month counseling induction: routine care (Active Comparator): Participants assigned to this condition will receive routine stepped-care treatment at ATS. Participants will begin in Step 2 (one counseling session per week), and be advanced to higher intensity care based on missed counseling sessions and drug-positive urine samples. Participants advanced to Step 3 will be scheduled to attend 2 group counseling sessions per week (in addition to individual counseling), and those advanced to Step 4 will be scheduled to attend 8 group counseling sessions per week (in addition to individual counseling). Time of methadone dosing will be based on step of care.
  Interventions: Behavioral: stepped-based care
- 3-month counseling induction: low threshold (Experimental): Participants assigned to this treatment arm will receive low threshold counseling. These participants will be scheduled to attend one counseling session per month with their individual counselor for the first 3-months. Participants can attend more counseling sessions if they desire, and they can meet with program supervisors to address crisis situations. They can receive methadone dosing any time during the clinic hours (7:30 am-1:15 pm and 4:00 pm - 6:00 pm)
  Interventions: Behavioral: low threshold care

INTERVENTIONS:
Behavioral: low threshold care — Low threshold care refers to a service delivery method that reduces the treatment demands for new admissions to substance abuse treatment. In the present study, participants will be scheduled to attend less counseling sessions, and will have greater access to methadone.
  Arms: 3-month counseling induction: low threshold
Behavioral: stepped-based care — Stepped-based care is routine treatment at ATS. Participants begin a low intensity care, and are advanced to more intensive levels of care (i.e., more intensive schedules of counseling) based on urine samples and counseling adherence.
  Arms: 3-month counseling induction: routine care

SUMMARY:
New admissions (n = 120) to the Addiction Treatment Services (ATS) will be stabilized on methadone and randomly assigned to one of two induction conditions: 1) routine stepped care, or 2) low threshold stepped care. All participants will continue with routine stepped care in month 4. Treatment retention is the primary outcome measure, while drug use (measured via weekly urinalysis testing) is the major secondary outcome.

DETAILED DESCRIPTION:
This randomized clinical trial will evaluate two induction strategies for helping out-of-treatment opioid abusers transition to methadone maintenance treatment. All study participants (n = 120) will be new admissions to the Addiction Treatment Services at Hopkins Bayview (ATS), stabilized on 80 mg of methadone, and randomly assigned to one of two study conditions. The experimental induction condition will receive low threshold stepped care (LTSC) for the first 3-month of treatment that reduces the counseling demands of maintenance treatment (i.e., one counseling session / month). This condition will be compared to routine stepped care (RSC) for the first 3-months, which provides escalating intensity of counseling schedules contingent on drug use or poor adherence. RSC is routine treatment at ATS. All participants will receive routine stepped care following the 3-month induction phase, and will have the opportunity to remain in treatment at ATS following study participation. Participation is for 4-months. Retention is the primary outcome. Participants will also submit urine samples weekly on a random schedule each month. We hypothesize that LTSC participants will exhibit better retention than RSC participants, and that both conditions will exhibit reductions in drug use compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* New admissions to methadone maintenance

Exclusion Criteria:

* Pregnant
* Acute medical or psychiatric condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
treatment retention | 120 days
  The number of days patients remained in treatment over the 120 day study.

SECONDARY OUTCOMES:
Drug use | weekly observation for 120 days
  Urinalysis testing is administered weekly, using a random testing schedule. Samples are tested for the presence of opioids, cocaine, and benzodiazepines

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Kidorf, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Addiction Treatment Services -- Hopkins Bayview, Baltimore, Maryland, United States